CLINICAL TRIAL: NCT01622192
Title: A Comparison Between the Repeatability of Probing Pocket Depths Achieved With Manual and Automated Periodontal Probes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH 16290
Record Dates: First submitted 2012-05-03; First posted 2012-06-19 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Disease
Keywords: Probing; manual probe; automated probe; Periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Automated probe (Experimental)
  Interventions: Device: Florida Probe automated probe

INTERVENTIONS:
Device: Florida Probe automated probe — Comparisons between the reproducibility of readings taken by an automated probe and a manual probe

SUMMARY:
The aim of the study is to determine the best method for measuring the extent and severity of the gum disease by comparing the repeatability of probing depths achieved by a manual probe when compared to an automated probe.

Hypothesis

The null hypothesis to be tested includes

* The automated probe does not improve the reproducibility of periodontal probing when compared to manual probing recordings
* The automated probe shows no advantage when comparing the reproducibility of

  * Moderate sites
  * Deep sites
  * Single vs. multirooted teeth
  * Different sextants
  * Different surfaces of teeth Buccal vs. palatal/lingual Mesial vs. mid vs. distal

DETAILED DESCRIPTION:
Measuring the clinical attachment loss using a periodontal probe is the benchmark by which attachment loss is diagnosed in periodontal disease. The accuracy and reproducibility of the probing measurements is an essential part of diagnosis, treatment planning and assessment of the treatment outcome. There are inherent errors associated with probing that have been identified in the literature. These relate to the operator technique, the probe used and the state of inflammation of the periodontal pocket/crevice.

The aim of this study is to compare the reproducibility of probing measurements using a probe tip with millimeter markings up to 15mm in the Florida probe ® handpiece. This tip will be used to allow conventional clinical measurements to be recorded at the same time as the electronic recordings on the Florida probe ®. The examiner would take the manual probe measurement and be blind to the electronic reading taken. The sites under question will have a second measurement recorded to allow assessment of the repeatability of the recordings. Therefore, from 2 probing passes 4 measurements would be obtained 2 manual and 2 electronic readings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Diagnosis of periodontitis (any form) but must have at least 2 sites in at least 1 sextant with a BPE code 4( pockets ≥ 5.5mm) at the time of screening
* Patient consent gained and has agreed to be a part of the study

Exclusion Criteria:

* Any medical condition that would exclude them from having the measurements taken
* Any medical problem that would make participation difficult
* If they do not have sufficient sites where probing depths are required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | pocket depth is reassessed at the same visit within 30 minutes
  Probing pocket depth with manual and electronic reading on single pass. Measurement repeated for one sextant.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth S Griffiths, BDS MRD FDS, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom